CLINICAL TRIAL: NCT07369921
Title: Comparison of Four Different Surgical Methods for the Treatment of Sacrococcygeal Pilonidal Sinus: a Randomized Controlled Trial
Brief Title: Pediatric Pilonidal Sinus Surgical Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zeliha Alicikus (Other Government)
Responsible Party: Sponsor-Investigator, Zeliha Alicikus, Assoc. prof. dr, Umraniye Education and Research Hospital
Organization: Umraniye Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z.AKIŞ
Record Dates: First submitted 2025-12-16; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Surgery; Pilonidal Sinus; Pediatric
Keywords: Pilonidal Sinus; pediatric surgery
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Intervention Model Description: randomized controlled
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Crystallized Phenol Applied Group (Group P) n:21 (Active Comparator): the pilonidal sinus (PS) periphery was cleaned using an antiseptic solution. A clamp was used to widen the sinus opening. The sinuses were thoroughly cleansed. Hair and granulation tissue were removed by curettage. Nitrofurantoin pomade (FurocinR Eczacıbaşı Istanbul, Turkey) was applied around the sinus to protect it from burns. Sufficient crystallized phenol (BotaFarma Medical Ankara, Turkey) was applied to fill the cavity (approximately 3-5 gr). Because crystallized phenol liquefies as soon as it contacts the body, it was compressed with a sponge for two minutes to prevent disintegration. The sinus opening was closed with ointment. Patients were hospitalized for one day.
  Interventions: Procedure: Crystallized Phenol Applied
- Endoscopy Group (Group EPSiT) n:22 (Active Comparator): The main sinus was enlarged to an initial width of 5 mm through which the pediatric cystoscope can pass. We utilized a 1% mannitol solution for sinus irrigation. The hair follicles and necrotic tissues were eliminated. Then, the sinus was effectively cauterized using a monopolar probe. The inside of the sinus was cleaned with a brush
  Interventions: Procedure: Crystallized Phenol Applied
- Limberg Flap Group (Group L) n:23 (Active Comparator): The sinus tract was marked with an iodine solution given through the sinus opening. The rhomboid shape was drawn with a sterile pen, with all sides being equal. The edges of the flap were sketched. the sinus area was completely removed, extending down to the presacral fascia. If iodine solution or sinus was seen outside the incision line, the excision area was enlarged to avoid residuals. The flap was released. A 10-French drainage catheter was inserted. Patients were discharged from the hospital on the third day after surgery.
  Interventions: Procedure: Crystallized Phenol Applied
- Modified Limberg Flap Group (Group ML) n:22 (Active Comparator): The sinus tract was marked with an iodine solution given through the sinus opening. The rhomboid shape was drawn with a sterile pen, with all sides being equal. The edges of the flap were sketched. the sinus area was completely removed, extending down to the presacral fascia. If iodine solution or sinus was seen outside the incision line, the excision area was enlarged to avoid residuals. The flap was released. A 10-French drainage catheter was inserted. Patients were discharged from the hospital on the third day after surgery.
  Interventions: Procedure: Crystallized Phenol Applied

INTERVENTIONS:
Procedure: Crystallized Phenol Applied — four different surgical methods for the treatment of sacrococcygeal pilonidal sinus
  Other Names: Endoscopy Group; Limberg Flap Group; Modified Limberg Flap Group

SUMMARY:
The aim of study to evaluate four different treatment options for pilonidal sinus disease in a randomized controlled trial to find the most suitable treatment option.

DETAILED DESCRIPTION:
Pilonidal sinus disease (PSD) is common in young adults and causes repeated infection and inflammation in the sacrococcygeal region. It is most common in men between the ages of 20 and 30, which is why most publications about PSD are part of adult series.

This study aims to determine which treatment option is more effective and beneficial for patients with sacrococcygeal pilonidal sinus. Furthermore, it aims to contribute to more positive treatment outcomes by identifying the causes of recurrence and morbidity in patients. Sacrococcygeal pilonidal sinus is quite common in adolescents. Treatment options vary from non-operative to endoscopic surgery. However, recurrence still occurs with every technique. Patients suffer from long treatment processes and morbidity. Although the exact causes of recurrence are not fully understood, it is thought that the patient's demographic characteristics and treatment option play a role. Most studies are retrospective and compare at most two treatment options. This is one of the reasons why it is not possible to reach a definitive conclusion about which treatment is more effective. Also, the number of studies conducted in the adolescent age group is limited. By conducting study prospectively and randomized, aim to prevent biased results.

ELIGIBILITY:
Inclusion Criteria:

* having sacrococcygeal pilonidal sinus disease
* written informed (family) consent were eligible for inclusion in this trial

Exclusion Criteria:

* Being over 18 years old or under 12 years old
* recurrent sacrococcygeal pilonidal sinus disease

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
complications | 30 days
  Recurrence
pain score | 24 hours
  VAS score under 4,VAS score above 4

SECONDARY OUTCOMES:
sinus volume measurement | 24 hours
  USG guided

CONTACTS AND LOCATIONS:
Locations (1):
- Umraniye Education and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No